CLINICAL TRIAL: NCT06716502
Title: A New Portable Device for PRE-hospital Non-invasive VENTilatory Support in Acute Respiratory Failure
Brief Title: A New Portable Device for Non-invasive Ventilatory Support
Acronym: PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Città di Lecce Hospital (Unknown)
Responsible Party: Principal Investigator, Giovanni Landoni, Director of the Research Center for Intensive Care and Anesthesiology of San Raffaele Scientific Institute, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-POC-2022-12376704
Record Dates: First submitted 2024-11-14; First posted 2024-12-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Respiratory Disease
Keywords: CPAP; NIV; Respiratory failure
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy elderly individuals (Experimental): The performance and easiness to use of the device will be evaluated in patients' self-experience conditions, with elderly participants self-applying the device.
  Interventions: Device: Portable CPAP usability assessment
- Patients with mild oxygenation impairment (Experimental): The efficacy of the device will be assessed in patients with mild oxygenation impairment.
  Interventions: Device: Portable CPAP efficacy

INTERVENTIONS:
Device: Portable CPAP efficacy — The device will be tested in providing a PEEP comprised between 4-7,5 cmH2O
  Arms: Patients with mild oxygenation impairment
Device: Portable CPAP usability assessment — The device usability will be evaluated in individual's self-experience tests, i.e., in conditions where the volunteer will self-apply the device.
  Arms: Healthy elderly individuals

SUMMARY:
Acute respiratory failure is a medical emergency rapidly leading to death, if not timely treated. Prompt Continuous Positive Airway Pressure (CPAP) improves patient outcomes. However, pre-hospital CPAP is currently limited to healthcare providers due to the absence of easy-to-use and immediate devices specifically designed for the non-medical population.

The efficacy and usability of a new portable CPAP device will be assessed. This device is specifically designed for potential use in out-of-hospital scenarios involving acute respiratory failure. The evaluation will focus not only on the performance of the device but also on its easiness of use.

DETAILED DESCRIPTION:
The efficacy and usability of a new portable CPAP device will be assessed in different clinical settings. The study will take place in three hospitals in Italy, with the objective of collecting data to support the future implementation of the device as a first-aid support tool for patients with respiratory failure in real-world scenarios.

ELIGIBILITY:
Arm 1

Inclusion Criteria:

1. Age ≥65 years
2. Clinically stable: non-hospitalized and not in acute illness
3. no professional medical knowledge: no experience as a health care provider
4. Ability to express informed consent as requested by the ethical committee

Arm 1 Exclusion Criteria: none

Arm 2

Inclusion Criteria:

1. Hospitalized adult patient
2. SpO2 of 90-93% in room air

Arm 2

Exclusion Criteria:

1. Facial burns/trauma/recent facial or upper airway surgery
2. Vomiting
3. Fixed upper airway obstruction
4. Undrained pneumothorax
5. Recent upper gastrointestinal surgery
6. Inability to protect the airway
7. Bowel obstruction
8. Patient refusal

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-19 (Estimated)

PRIMARY OUTCOMES:
Device easiness-to-use | Up to 2 hours
  Volunteers in self-experience tests will be asked to assign a score depending on the easiness-to-use of the device and comfort during the device operation.
  A semantic differential scale will be used between "hard to use" (corresponding to the score 1) and "easy to use" (corresponding to the score 5). The best result is represented by a higher score, with 5 being the highest and 1 the lowest.
Duration of proper pressure delivery | Up to 2 hours
  Total time of target pressure (4 - 15 cmH2O) during 15-min test
Battery power consumption and duration | Up to 2 hours
  We will set 15 minutes of continuous device operation as an efficacy threshold and will assess the battery status at the end of each experiment.
Change in SpO2 level | Up to 2 hours
  Change in SpO2 before and during the device application

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Study Chair — IRCCS San Raffaele
Locations (3):
- Italy (3):
  - Città di Lecce Hospital, Lecce, Apulia
  - IRCCS San Raffaele, Milan
  - Università degli studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: No